CLINICAL TRIAL: NCT01802801
Title: Intra-and Inter-observer Agreement in the Morphological Assessment of Human Embryos
Brief Title: Intra- and Interobserver Agreement in the Assessment of Human Embryos
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Prof. Dr., University Hospital, Gasthuisberg
Other Study IDs: GP12122007
Record Dates: First submitted 2010-03-25; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: the Focus of This Study is to Measure the Intra- and Interobserver Agreement for the Evaluation of Early Stage Embryos
MeSH Terms: interventions — Embryonic Development

GROUPS / COHORTS (1):
- 1
  Interventions: Other: embryo development

INTERVENTIONS:
Other: embryo development — intra- and inter-observator analysis

SUMMARY:
The purpose of this study is to determine the intra- and interobserver agreement.

ELIGIBILITY:
Inclusion Criteria:

* fertilized embryos

Exclusion Criteria:

* unfertilized embryos

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: embryos of IVF/ICSI patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the intra- and inter-observer variability in the assessement of human embryos
  Variation in observer assessment of embryo characteristics on day 1, 2 and 3 of embryo development. Assessment of these characteristics is standard procedure. Safety and tolerability or efficacy issues are not relevant for this outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Catholic University Leuven, Leuven, Belgium